CLINICAL TRIAL: NCT04803201
Title: A Randomized Phase II Study of CHO(E)P vs CC-486-CHO(E)P vs Duvelisib-CHO(E)P in Previously Untreated CD30 Negative Peripheral T-Cell Lymphomas
Brief Title: Testing the Addition of Duvelisib or CC-486 to the Usual Treatment for Peripheral T-Cell Lymphoma
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim Analysis
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A051902; NCI-2021-01380 (Registry Identifier: NCI Clinical Trial Reporting Program); U10CA180821 (NIH)
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Angioimmunoblastic T-cell Lymphoma; Enteropathy-Associated T-Cell Lymphoma; Follicular T-Cell Lymphoma; Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Monomorphic Epitheliotropic Intestinal T-Cell Lymphoma; Nodal Peripheral T-Cell Lymphoma With TFH Phenotype; Peripheral T-Cell Lymphoma, Not Otherwise Specified
MeSH Terms: conditions — Immunoblastic Lymphadenopathy; Enteropathy-Associated T-Cell Lymphoma; Lymphoma, T-Cell | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Etoposide; duvelisib; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (duvelisib, CHO[E]P) (Experimental): Patients receive cyclophosphamide IV on day 1, doxorubicin IV on day 1, vincristine IV on day 1, etoposide IV on day 1 or days 1-3 or PO QD on days 2-3 for patients =< 60 years old, and prednisone PO QD on days 1-5. Patients also receive duvelisib PO BID on days 1-21. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Etoposide; Drug: Duvelisib
- Arm B (CC-486, CHO[E]P) (Experimental): Patients receive cyclophosphamide IV on day 1, doxorubicin IV on day 1, vincristine IV on day 1, etoposide IV on day 1 or days 1-3 or PO QD on days 2-3 for patients =< 60 years old, and prednisone PO QD on days 1-5. Patients also receive CC-486 PO QD on days -6 to 0 of cycle -1 and days 8-21 of cycles 1-5. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Etoposide; Drug: Oral azacitidine
- Arm C (CHO[E]P) (Active Comparator): Patients receive cyclophosphamide IV on day 1, doxorubicin IV on day 1, vincristine IV on day 1, etoposide IV on day 1 or days 1-3 or PO QD on days 2-3 for patients =< 60 years old, and prednisone PO QD on days 1-5. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Etoposide

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
Drug: Doxorubicin — Given IV
Drug: Vincristine — Given IV
Drug: Prednisone — Given PO
Drug: Etoposide — Given IV or PO
Drug: Duvelisib — Given PO
  Arms: Arm A (duvelisib, CHO[E]P)
Drug: Oral azacitidine — Given PO
  Arms: Arm B (CC-486, CHO[E]P)

SUMMARY:
This phase II trial studies the effect of duvelisib or CC-486 and usual chemotherapy consisting of cyclophosphamide, doxorubicin, vincristine, etoposide, and prednisone in treating patients with peripheral T-cell lymphoma. Duvelisib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as CC-486, cyclophosphamide, doxorubicin, vincristine, etoposide and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. This trial may help find out if this approach is better or worse than the usual approach for treating peripheral T-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the complete remission (CR) rates by positron emission tomography (PET)/computed tomography (CT) following completion of treatment with duvelisib-cyclophosphamide (C) doxorubicin (H) vincristine (O) (etoposide [E]) prednisone (P) versus (vs) CHO(E)P and with oral azacitidine (CC-486)-CHO(E)P vs CHO(E)P in previously untreated peripheral T-cell lymphomas that have < 10% expression of CD30.

SECONDARY OBJECTIVES:

I. To determine the toxicity and tolerability of the treatment regimens. II. To determine the overall response rate (ORR), duration of response, progression free survival (PFS), event free survival (EFS), and overall survival (OS) of each treatment regimen.

III. To determine whether designation of follicular helper T-cell phenotype is correlated with response to therapy, PFS, EFS, and OS.

IV. To assess the toxicity profile of the experimental regimens in untreated CD30 negative peripheral T-cell lymphomas using Common Terminology Criteria for Adverse Events (CTCAE) and patient reported outcomes (PRO)-CTCAE.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM A: Patients receive cyclophosphamide intravenously (IV) on day 1, doxorubicin IV on day 1, vincristine IV on day 1, etoposide IV on days 1-3 or etoposide IV on day 1 and orally (PO) once daily (QD) on days 2-3 for patients <=60 years old, and prednisone PO QD on days 1-5. Patients also receive duvelisib PO twice daily (BID) on days 1-21. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive cyclophosphamide IV on day 1, doxorubicin IV on day 1, vincristine IV on day 1, etoposide IV on days 1-3 or etoposide IV on day 1 and orally (PO) once daily (QD) on days 2-3 for patients <=60 years old, and prednisone PO QD on days 1-5. Patients also receive CC-486 PO QD on days -6 to 0 of cycle -1 and days 8-21 of cycles 1-5. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive cyclophosphamide IV on day 1, doxorubicin IV on day 1, vincristine IV on day 1, etoposide IV on days 1-3 or etoposide IV on day 1 and orally (PO) once daily (QD) on days 2-3 for patients <=60 years old, and prednisone PO QD on days 1-5. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 6 weeks after cycle 6 day 1, then every 12 weeks for 2 years, then every 24 weeks until 5 years from end of treatment or until documented progression of lymphoma. After documented progression of lymphoma, patients are followed up every 6 months until 5 years from end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of peripheral T-cell lymphoma (PTCL) with < 10% CD30 expression by immunohistochemistry in the following subtypes (by local review): nodal T-cell lymphoma with T-follicular helper (TFH) phenotype (TFH-PTCL), follicular T-cell lymphoma, PTCL-not otherwise specified (NOS), angioimmunoblastic T-cell lymphoma (AITL), enteropathy associated T-cell lymphoma, monomorphic epitheliotropic intestinal T-cell lymphoma

  * Patients with expression of CD30 in >= 10% of the tumor (based on local immunohistochemistry review) regardless of histology will not be permitted
  * Patients with a diagnosis of other PTCL subtype histologies other than those specified in the inclusion criteria are excluded including large cell transformation of mycosis fungoides
  * Patients will be stratified by presence or absence of TFH phenotype (i.e. diagnosis of AITL, TFH-PTCL, follicular T-cell lymphoma) based on local review of pathology. Determination of TFH phenotype can be defined by expression of two or more of the following markers CD10, BCL6, CXCL13, ICOS, and PD1 by immunohistochemistry
* Measurable disease as defined by the Lugano criteria
* No prior systemic therapy for lymphoma (excluding corticosteroids)
* Not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown. Therefore, for women of childbearing potential only, a negative urine or serum pregnancy test done =< 7 days prior to registration is required
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Platelet count >= 75,000/mm^3 (>= 50,000/mm^3 if secondary to bone marrow involvement from lymphoma per investigator assessment; the first 12 patients on each arm of the study must have platelets >= 75,000/mm^3 regardless of bone marrow involvement)
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) or alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) =< 3.0 x upper limit of normal (ULN)

  * Except in subjects with documented liver involvement by lymphoma
* Calculated creatinine clearance >= 30 mL/min by Cockcroft-Gault formula
* Total bilirubin =< 2.0 x ULN

  * Except in cases of Gilbert's Syndrome or documented liver or pancreatic involvement by lymphoma
* Archival tissue must be available for submission
* Patients known to have HTLV 1/2 are excluded
* Patients with known central nervous system involvement are excluded
* No active viral infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C. Those who are seropositive (e.g. hepatitis B core antibody [Ab] positive) are permitted if they are negative by polymerase chain reaction (PCR). Those who are seropositive for hepatitis B and are negative for hepatitis B virus (HBV) deoxyribonucleic acid (DNA) by PCR must receive concomitant hepatitis B directed antiviral therapy. Those who have hepatitis C Ab positivity who have completed curative therapy for hepatitis C with negative hepatitis C PCR are eligible
* Patients with history of HIV are eligible if they have an undetectable viral load for at least 6 months
* No active uncontrolled systemic fungal, bacterial or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy and/or other treatment). Patients with Epstein-Barr virus (EBV) viremia related to their lymphoma are permitted
* No concurrent malignancy requiring active therapy within the last 3 years with the exception of basal cell carcinoma limited to the skin, squamous cell carcinoma limited to the skin, carcinoma in situ of the cervix, breast or localized prostate cancer. Adjuvant hormonal therapy for cancer previously treated for curative intent is permitted
* Patients must have documented left ventricular ejection fraction of >= 45%
* No significant active cardiac disease within the previous 6 months including:

  * New York Heart Association (NYHA) class III or IV congestive heart failure
  * Unstable angina or angina requiring surgical or medical intervention; and/or
  * Myocardial infarction
* No contraindication to any drug in the chemotherapy regimen, including neuropathy >= grade 2
* Chronic concomitant treatment with strong inhibitors of CYP3A4 is not allowed on this study. Patients on strong CYP3A4 inhibitors must discontinue the drug for 14 days prior to registration on the study. Chronic concomitant treatment with strong CYP3A4 inducers is not allowed. Patients must discontinue the drug 14 days prior to the start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete remission (CR) rate | Up to 6 months
  Defined as the number of patients with complete remission (CR) divided by the total number of patients randomized. Will be measured by fludeoxyglucose F-18 (FDG) positron emission tomography (PET)/computed tomography (CT) at the completion of treatment (at end of treatment) and will be compared between each experimental arm and control arm. Final analyses will use z-scores obtained from a stratified Cochran-Mantel-Haenszel test to compare the CR rates between each experimental arm and control arm. For each treatment arm, CR rates will be estimated with their 95% confidence intervals.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 5 years
  Adverse events will be collected and graded according to the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 criteria. For CTCAE data, the maximum grade for each type of adverse will be recorded for each patient, and described using frequency tables. All-cause adverse events will be summarized as well as treatment-related adverse events.
Overall response rate (ORR) | Up to 6 months
  Overall response includes complete and partial remissions by FDG PET/CT at the completion of treatment (at end of treatment). ORR will be estimated for each treatment arm and calculated as the number of patients with response divided by the total number of patients randomized. For each treatment arm, ORRs will be estimated with their 95% confidence intervals. ORR at the interim assessment will be summarized in the same manner, and how response changes between the interim and final assessment will be described.
Duration of response | From first date of complete or partial remission until the earlier of disease progression, death from any cause, or non-protocol lymphoma-directed therapy to treat residual or progressive disease, assessed up to 5 years
  The Kaplan-Meier method will be used to estimate duration of response for each treatment arm, with 2-year estimates and medians along with their 95% confidence intervals.
Progression-free Survival (PFS) | From randomization date until the earlier of disease progression, death from any cause, or non-protocol lymphoma-directed therapy to treat residual or progressive disease, assessed up to 5 years
  The Kaplan-Meier method will be used to estimate PFS for each treatment arm, with 2-year PFS estimates and PFS medians along with their 95% confidence intervals.
Event-free Survival (EFS) | From randomization date until earlier of non-protocol lymphoma-directed therapy for any reason (excluding planned consolidative transplant), disease progression, or death from any cause, assessed up to 5 years
  The Kaplan-Meier method will be used to estimate event-free survival (EFS) for each treatment arm, with 2-year EFS estimates and EFS medians along with their 95% confidence intervals.
Overall Survival (OS) | From randomization date until death from any cause, censoring patients alive at the date of last contact, assessed up to 5 years
  The Kaplan-Meier method will be used to estimate overall survival (OS) for each treatment arm, with 2-year OS estimates and OS medians along with their 95% confidence intervals.
Correlation of follicular helper T-cell phenotype with response, PFS, EFS and OS | Up to 5 years
  CR rates and ORRs will be estimated with 95% confidence intervals for patients with and without the follicular helper T-cell phenotype, as well for patients with the peripheral T-cell lymphomas (PTCL) genotype.
Patient reported outcomes (PROs) | Up to 6 months
  Patient reported outcomes (PROs) will be captured using the NCI PRO-CTCAE. Scores (0-4) and maximum score for each PRO-CTCAE item, with and without taking into account whether it is worse than the patient's own baseline score, will be recorded for each patient. PRO-CTCAE data will, at minimum, be analyzed similarly to CTCAE data.

CONTACTS AND LOCATIONS:
Overall Officials: Neha Mehta-Shah, MD, MSCI, Study Chair — Washington University School of Medicine
Locations (86):
- United States (86):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Miami Valley Hospital South, Centerville, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin